CLINICAL TRIAL: NCT07313605
Title: Beta-Blocker Therapy Versus Standard Care in Patients With Septic Shock: A Pilot Randomized Controlled Trial Utilizing Predictive Enrichment With Point-of-Care Ultrasound
Brief Title: POCUS-Guided Esmolol in Septic Shock: A Pilot RCT
Acronym: Epic-Beta
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Basmaji (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Western University, Canada (Other)
Responsible Party: Sponsor-Investigator, John Basmaji, "Assistant Professor, Division of Critical Care Medicine, Department of Medicine, Western University, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 127880
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Patients randomized to this arm will receive standard care for septic shock according to Surviving Sepsis Campaign guidelines. This includes fluid resuscitation, a mean arterial pressure target of 65 mmHg or greater, early broad-spectrum antibiotics, source control when applicable, vasopressor support with norepinephrine as the first-line agent, stress-dose corticosteroids, early nutrition, and lung-protective mechanical ventilation when required. Beta-blockers and calcium channel blockers are prohibited throughout the 5-day study period. For patients who develop new-onset atrial fibrillation or flutter, amiodarone will be the preferred first-line antiarrhythmic agent. Treating physicians may use other antiarrhythmic medications at their discretion, provided they are not beta-blockers or calcium channel blockers.
- Esmolol (Experimental): Patients will receive an intravenous infusion of esmolol, an ultra-short-acting cardioselective beta-1 adrenergic receptor antagonist with a half-life of approximately 9 minutes. The infusion will be titrated to achieve a target heart rate of 75-95 beats per minute, with a maximum dose of 300 mcg/kg/minute. Treatment will continue for a maximum of 5 days or until ICU discharge, death, or resolution of shock (defined as discontinuation of vasopressors for at least 6 hours). Esmolol will be the preferred first-line treatment for tachyarrhythmias. All patients will continue to receive standard care for septic shock per Surviving Sepsis Campaign guidelines.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — Patients will receive an intravenous infusion of esmolol, an ultra-short-acting cardioselective beta-1 adrenergic receptor antagonist with a half-life of approximately 9 minutes. The infusion will be titrated to achieve a target heart rate of 75-95 beats per minute, with a maximum dose of 300 mcg/kg/minute. Treatment will continue for a maximum of 5 days or until ICU discharge, death, or resolution of shock (defined as discontinuation of vasopressors for at least 6 hours). Esmolol will be the preferred first-line treatment for tachyarrhythmias. All patients will continue to receive standard care for septic shock per Surviving Sepsis Campaign guidelines.
  Arms: Esmolol

SUMMARY:
The goal of this pilot clinical trial is to determine if conducting a larger study using point-of-care ultrasound (POCUS) to guide beta-blocker therapy in patients with septic shock is feasible. Septic shock is a life-threatening condition where infection causes dangerously low blood pressure, requiring medications to support the heart and circulation. In septic shock, the body's stress response causes the heart to beat too fast, which can worsen organ damage.

Beta-blockers are medications that slow the heart rate and may improve outcomes, but previous studies have shown mixed results. Some patients may be harmed by beta-blockers if they have not received enough fluids or if their heart is not functioning well. This study uses ultrasound to identify patients who are most likely to benefit and least likely to be harmed by beta-blocker therapy.

The main questions this study aims to answer are: Is it feasible to recruit patients, obtain consent, perform ultrasound screening, and follow the study protocol? Researchers will compare two groups: one receiving the beta-blocker esmolol versus another receiving standard care, to assess the feasibility of a larger trial.

Participants in the esmolol group will receive an intravenous infusion titrated to achieve a target heart rate of 75-95 beats per minute for up to 5 days or until shock resolves. All participants will be monitored for 90 days to track survival and organ function.

DETAILED DESCRIPTION:
Septic shock remains a leading cause of intensive care unit admissions and mortality worldwide, with approximately 50% of affected patients dying. Excess beta-adrenergic activity, triggered by the body's stress response, drives much of this mortality by causing persistent tachycardia, increased myocardial oxygen consumption, reduced coronary perfusion, impaired cardiac output, endothelial dysfunction, and cellular metabolic derangements.

Beta-adrenergic blockers offer a physiologically plausible approach to counteract these harmful effects. A meta-analysis of 12 randomized controlled trials enrolling 1170 patients suggests beta-blockers may reduce 28-day mortality (risk ratio 0.76, 95% confidence interval 0.62-0.93). However, substantial heterogeneity exists across trials, with results ranging from a 44% mortality reduction to an 11% increase. One multicenter trial was stopped early for potential harm. This heterogeneity may be explained by inadvertent enrollment of patients at high risk of harm from beta-blockade: those with inadequate fluid resuscitation who depend on tachycardia to maintain cardiac output, and those with left or right ventricular dysfunction who cannot tolerate the negative inotropic effects of beta-blockers.

This pilot trial implements a predictive enrichment strategy using point-of-care ultrasound to exclude high-risk phenotypes before randomization. Eligible patients undergo POCUS assessment of fluid responsiveness using left ventricular outflow tract velocity time integral or carotid corrected flow time with passive leg raise. Patients demonstrating fluid responsiveness (greater than 15% change) are excluded as inadequately resuscitated. Cardiac function assessment excludes patients with moderate to severe left ventricular systolic dysfunction (ejection fraction less than 35%) or right ventricular dysfunction (tricuspid annular plane systolic excursion less than 17mm, severe RV dilation, septal shift, or RV S prime less than 9.5 cm/second).

Patients meeting eligibility criteria after POCUS screening are randomized 1:1 to esmolol or standard care. The intervention arm receives intravenous esmolol initiated at 50 mcg/kg/minute and titrated by 50 mcg/kg/minute every 15 minutes to achieve a target heart rate of 75-95 beats per minute, with a maximum dose of 300 mcg/kg/minute. Treatment continues for up to 5 days or until ICU discharge, death, or discontinuation of vasopressors for at least 6 hours. Both arms receive standard septic shock management per Surviving Sepsis Campaign guidelines.

Primary outcomes focus on feasibility: recruitment rate (target 4 patients per month), consent rate (target 80% or greater), POCUS screening completion rate (target 80% or greater), and protocol adherence (target 80% or greater). Secondary outcomes include 28-day and 90-day mortality, days alive and free of organ support therapies, and ICU and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Within 24 hours of diagnosis of septic shock based on Sepsis-3 criteria (requirement for vasopressors to maintain organ perfusion, lactate greater than 2 mmol/L, suspected or confirmed infection)
3. Within 72 hours of ICU admission
4. Tachycardia with heart rate 100 beats per minute or greater, defined as either sinus tachycardia or atrial fibrillation/flutter

Exclusion Criteria:

1. Known allergy to beta-blockers
2. Second or third-degree heart block without a functioning pacemaker
3. Acute bronchospasm or status asthmaticus
4. Pregnancy
5. Patient receiving extracorporeal membrane oxygenation
6. Decision to limit life-sustaining therapies
7. Untreated pheochromocytoma
8. Fluid-responsive patients as determined by POCUS assessment
9. Moderate to severe right ventricular and/or systolic left ventricular dysfunction as determined by POCUS assessment
10. Patient already receiving calcium channel blocker or beta-blocker therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From study initiation to end of recruitment, approximately 25 months
  Number of participants enrolled during the recruitment period who successfully complete study procedures and follow-up.
Consent Rate | From study initiation to end of recruitment, approximately 25 months
  The total number of eligible participants consented divided by the total number of eligible participants approached for consent
POCUS Screening Completion Rate | From study initiation to end of recruitment, approximately 25 months
  Number of participants who successfully underwent fluid responsiveness and cardiac function evaluation using point-of-care ultrasound, divided by the total number of participants eligible for POCUS screening. A successful POCUS entails acquiring adequate quality images for interpretation and providing conclusive assessments of fluid responsiveness, left ventricular function, and right ventricular function.
Protocol Adherence | From day of randomization (day 1) to day 5
  Intervention arm: The number of participants who received esmolol as per protocol divided by the total number of participants randomized to the intervention arm, and the total time spent within heart rate target divided by total time on esmolol infusion. Control arm: The number of participants who did not receive any beta-blocker therapy during the 5-day study period divided by the total number randomized to the control arm.

SECONDARY OUTCOMES:
28-Day Mortality | From randomization to 28 days
90-Day Mortality | From randomization to 90 days
Duration of Mechanical Ventilation | From randomization to 28 days
Duration of Vasoactive Medications | From randomization to 28 days
Provision of Renal Replacement Therapy | From randomization to 28 days

OTHER OUTCOMES:
Heart Rate Separation | From randomization to day 5
Mean Arterial Pressure | From randomization to day 5
Vasopressor Requirements | From randomization to day 5
Bradycardia Episodes | From randomization to day 5
Bradycardia Episodes Requiring Intervention | From randomization to day 5
Hypotension Episodes | From randomization to day 5
Hypotension Episodes Requiring Intervention | From randomization to day 5
Cardiac Complications | From randomization to day 5
  New-onset arrhythmias, second or third degree heart block, or cardiogenic shock
Serious Adverse Events | From randomization to day 5
  Any adverse event that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening, or results in death.

CONTACTS AND LOCATIONS:
Overall Officials: John Basmaji, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McChesney C, Orozco N, Fiorini K, Wong MYS, Slessarev M, Prager R, Kao R, Leligdowicz A, Sharif S, Lewis K, Rochwerg B, Honarmand K, Ball IM, Arntfield R, Houlton R, VanNynatten L, Basmaji J. Impact of Short-Acting Beta-Blockers on the Outcomes of Patients With Septic Shock: A Systematic Review and Meta-Analysis. Crit Care Med. 2025 May 1;53(5):e1125-e1139. doi: 10.1097/CCM.0000000000006604. Epub 2025 Feb 26. PMID 40009025